CLINICAL TRIAL: NCT00826865
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Levetiracetam 750 mg Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of Levetiracetam 750 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LEVE-T750-PVFS-1
Record Dates: First submitted 2009-01-15; First posted 2009-01-22 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam — 750 mg tablet
  Other Names: KEPPRA

SUMMARY:
The objective of this study was to prove the bioequivalence of Levetiracetam 750 mg Tablets under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to Levetiracetam or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
bioequivalance based on Cmax | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allison, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States